CLINICAL TRIAL: NCT00921414
Title: Manteau 2007 SJ "LYMA" "Randomized, Open-label, Phase III Study Efficacy of Rituximab Maintenance Therapy in Patients 18 to 65 Years , First-line Treatment for MCL
Brief Title: Mantel Cell Lymphoma Efficacy of Rituximab Maintenance
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French Innovative Leukemia Organisation (Other)
Collaborators: Lymphoma Study Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Manteau 2007 SJ "LYMA"
Record Dates: First submitted 2009-05-27; First posted 2009-06-16 (Estimated); Last update posted 2018-04-27 (Actual); Status verified 2018-04

CONDITIONS: Mantle Cell Lymphoma
Keywords: Mantle cell lymphoma; R DHAP; ASCT; Rituximab Maintenance
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Rituximab; Observation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): observation : 3 years maintenance period with assesments and surveillance every 2 months
  Interventions: Other: Watch and wait
- 2 (Experimental): maintenance period infusions of Rituximab 375 mg/m2/2 months and assessement and surveillance
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 2 months after ASCT maintenance treatment with Rituximab 500mg/m² IV every 2 months during 3 years
  Other Names: Mabthera®
  Arms: 2
Other: Watch and wait — No treatment patient follow-up every 2 months during 3 years
  Other Names: observation
  Arms: 1

SUMMARY:
Randomized, open-label, phase III study to evaluate the efficacy of rituximab maintenance therapy in patients aged between 18 and 65 years inclusive undergoing first-line treatment for mantle cell lymphoma and exhibiting a response after autologous transplantation.

DETAILED DESCRIPTION:
Demonstration of the superiority in terms of 4-year event-free survival (EFS) of Rituximab maintenance therapy compared to post-autograft surveillance in patients aged 18-65 years inclusive, treated with R-DHAP then autologous transplantation for MCL as first-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* mantle cell lymphoma
* Initial immunophenotyping with CD20 and CD5.
* CD20+.
* t (11;14) by karyote, FISH, molecular biology or immunohistochemistry (Bcl-1)
* Patient no previous treated.
* At least one tumor site accessible for assessment
* Aged > 18 years < 65
* ECOG < or = 2.
* No other neoplasms apart from resected basal cell carcinoma or in situ carcinoma.
* signed informed consent
* FEVG 50%

Exclusion Criteria:

* other type of lymphoma
* ECOG > or = 3
* relapse
* serology VIH + Hepatite +
* diabetis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2008-09; Primary Completion 2008-09 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
event-free survival (EFS) post Rituximab maintenance therapy | EFS post 4 years after maintenance

SECONDARY OUTCOMES:
duration of PFS of the entire group of patients. | Safety/efficacy of maintenance treatment
duration of OS of the entire group of patients | safety/efficacy of treatment
complete, partial and overall response rate after induction with R-DHAP and after ASCT. | safety/efficacy of all the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Steven LE GOUILL, MD, Principal Investigator — French Innovative Leukemia Organisation
Locations (1):
- Regional University Hospital, Nantes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sarkozy C, Callanan M, Thieblemont C, Oberic L, Burroni B, Bouabdallah K, Damaj G, Tessoulin B, Ribrag V, Houot R, Morschhauser F, Griolet S, Joubert C, Cacheux V, Delwail V, Safar V, Gressin R, Cheminant M, Delfau-Larue MH, Hermine O, Macintyre E, Le Gouill S. Obinutuzumab vs rituximab for transplant-eligible patients with mantle cell lymphoma. Blood. 2024 Jul 18;144(3):262-271. doi: 10.1182/blood.2024023944. PMID 38669626
- [Derived] Le Gouill S, Thieblemont C, Oberic L, Moreau A, Bouabdallah K, Dartigeas C, Damaj G, Gastinne T, Ribrag V, Feugier P, Casasnovas O, Zerazhi H, Haioun C, Maisonneuve H, Houot R, Jardin F, Van Den Neste E, Tournilhac O, Le Du K, Morschhauser F, Cartron G, Fornecker LM, Canioni D, Callanan M, Bene MC, Salles G, Tilly H, Lamy T, Gressin R, Hermine O; LYSA Group. Rituximab after Autologous Stem-Cell Transplantation in Mantle-Cell Lymphoma. N Engl J Med. 2017 Sep 28;377(13):1250-1260. doi: 10.1056/NEJMoa1701769. PMID 28953447
- See also: FILO Website — http://www.filo-leucemie.org